CLINICAL TRIAL: NCT01358617
Title: Observational - Expression of Ubiquitin Carboxyl-Terminal Hydrolase 1 (UCHL1) in Neuroblastoma Cancer Stem Cells and Its Relationship to Patient Prognosis
Brief Title: Prognostic Biomarkers in Tumor Tissue Samples From Young Patients With Neuroblastoma
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ANBL11B3; NCI-2011-02856 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); U10CA098543 (NIH)
Record Dates: First submitted 2011-05-19; First posted 2011-05-23 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Disseminated Neuroblastoma; Localized Resectable Neuroblastoma; Localized Unresectable Neuroblastoma; Recurrent Neuroblastoma; Stage 4S Neuroblastoma
MeSH Terms: conditions — Neuroblastoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Tumor Tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Biomarker analysis: Archived tissue microarray samples are analyzed for ubiquitin carboxyl-terminal hydrolase 1 (UCHL1) expression by UCHL1 monoclonal antibody and peroxidase technique.
  Interventions: Other: diagnostic laboratory biomarker analysis

INTERVENTIONS:
Other: diagnostic laboratory biomarker analysis — Correlative studies

SUMMARY:
This research study is studying biomarkers in tumor tissue samples from young patients with neuroblastoma. Studying samples of tissue from patients with cancer in the laboratory may help doctors identify biomarkers and learn more about biomarkers related to cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine whether ubiquitin carboxyl-terminal hydrolase 1 (UCHL1) expression is an indirect cancer stem cell marker in pediatric patients with neuroblastoma. Correlate UCHL1 expression with staging information and patient's outcome.

Study Subtype: Observational Observational Study Model: Case-control Time Perspective: Retrospective Biospecimen Retention: None Retained Biospecimen Description: Tissue Study Population Description: Tissue microarray samples from patients with Neuroblastoma supplied by the COG Biopathology Center Sampling Method: Probability

OUTLINE:

Archived tissue microarray samples are analyzed for ubiquitin carboxyl-terminal hydrolase 1 (UCHL1) expression by UCHL1 monoclonal antibody and peroxidase technique. Results are then compared with patients' clinical data, including age at diagnosis, race, date of diagnosis, histology, stage and location at diagnosis, presence of cancer predisposition, date of completion of treatment, surgery performed, type of chemotherapy received, history of recurrence, and status (alive with disease, alive without disease, dead), if available.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with neuroblastoma
* Tissue microarrays containing normal and neuroblastoma samples provided by the Children's Oncology Group (COG) Biopathology Center

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients With Neuroblastoma
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2011-05; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Association between test result (percent cells with positive UCHL1 staining dichotomized into high and low categories) and International Neuroblastoma Staging System (INSS) stage | Baseline

SECONDARY OUTCOMES:
Relationship between UCHL1 expression and tumor histology, and MYCN amplification | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Sugalski, MD, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Monrovia, California, United States